CLINICAL TRIAL: NCT00375063
Title: Prospective Randomized Study of Unprotected Left Main Stenting Versus Bypass Surgery
Brief Title: Study of Unprotected Left Main Stenting Versus Bypass Surgery (LE MANS Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ministry of Science and Higher Education, Poland (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6 P05B 132 21
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-09

CONDITIONS: Coronary Artery Stenosis; Myocardial Revascularization; Myocardial Ischemia
Keywords: left main stenosis; Percutaneous Coronary Intervention; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Coronary Stenosis; Myocardial Ischemia | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention
Procedure: Coronary Artery Bypass Grafting

SUMMARY:
Unprotected left main coronary artery (ULMCA) stenting, offering restoration of a native flow to left coronary artery, is the subject of intense investigations as a potential alternative to bypass surgery. The purpose of the study is to compare the short and long term results of unprotected left main stenting with coronary artery bypass surgery.

DETAILED DESCRIPTION:
The natural history and the results of pharmacological treatment in patients with severe narrowing of left main coronary artery show very poor prognosis (5 year survival less than 50%).

There is general agreement that surgical treatment improves 5 year survival in patients with left main coronary artery obstruction 3, however long term survival rate (15 year follow-up) is low in both groups (37% and 27% respectively in surgical and medical group). Median survival was longer in surgical group in general population (13.3 vs 6.6 years) , but there was no significant difference in patients with normal LV ejection fraction (14.7 vs 15 years).

With the advent of coronary stenting encouraging results were reported by several authors. There was high success rate 98-100% for elective procedures and in these series the mortality (for protected and non-protected left main) ranged from 0 to 3.4 %, and 6 month event free survival rate was 70-80%. Restenosis rate in stented LM varied from 10-22% for proximal LM to 40% for distal LM. Final minimal luminal area >=7mm2 post procedure, assessed by IVUS, predicted low restenosis rate of 7%, while the area below <7mm2 was connected with restenosis of 50%. Our and other experience showed that left main in-stent restenosis can be treated successfully with another percutaneous intervention (including endarterectomy and balloon angioplasty) as well as by surgical revascularization.

Six and 12-month survival rate depended on the LV function. Patients with LVEF>40% had in-hospital event free survival of 98% and 9-month event free survival of 86%, whereas patients with LVEF <40% had in-hospital and 9 month event-free survival of 67 and 22% respectively. Additionally, in patients presented with acute myocardial infarction or bail-out procedures, early and late results of LM stenting were not as good as for elective cases.

Our previously presented promising results of left main stenting is mainly related to proper technique of LM stenting (short inflations within LM, careful guiding catheter manipulation, stent selection), as well as very cautiously designed follow-up (every month visit for first six month, routine coronary angiography within 3-6 months after procedure). This initial experience gives us the backgrounds for a larger prospective randomized trial comparing elective surgical revascularisation and percutaneous intervention in patients with LM coronary artery disease. It is our impression that design and the delivery system of the new generation stent is uniquely suited to safely treat this difficult subset of patients. At the present time we would limit the study to the discrete lesions in proximal (ostial and mid) left main with reference luminal diameter >=3 mm. Based on published results of stenting under IVUS examination for such a lesion we estimate the restenosis rate to be well below 10%. As we expect, the survival and complication rate within one year in both group will be similar. Therefore our main concern is weather both treatment strategies will offer the same prevention of LV function, as well as improvement of functional capacity and coronary reserve in both groups in a period of 2-3 years.

ELIGIBILITY:
Inclusion Criteria:

* The patients' age 18 to 80
* Significant LM stenosis (>50%)
* The target vessel reference diameter 2.5mm.
* Concomitant multivessel disease suitable for PCI is allowed.
* The patient is an acceptable candidate for coronary artery bypass surgery.
* The patient agreement for 6 month follow-up cardiac catheterization, which will include left ventricular angiogram.
* The patient written informed consent.

Exclusion Criteria:

* An allergy or contraindication to aspirin, ticlopidine or Clopidogrel.
* Presence of diffuse, significant (>++) calcifications in LM
* Left ventricular ejection fraction < 35%
* History of bleeding diathesis or coagulopathy.
* Any previous PCI or CABG surgery
* Acute MI within 48 hours, cardiogenic shock.
* Bail-out stenting of dissected LM during complicated PCI.
* The patient suffered a stroke or transient ischemic neurological attack (TIA) within 3 months.
* Chronic renal insufficiency.
* Positive pregnancy test.
* Any disease that may shorten the life expectancy of the patient.
* The patient is currently participating in another research study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2001-01; Study Completion 2005-12

PRIMARY OUTCOMES:
LV function assessed by 2D echocardiography
exercise tolerance measured with ECG treadmill stress testing
angina severity according to CCS classification 12 months after the index intervention

SECONDARY OUTCOMES:
30 day and one year major adverse events (MAE)
30 day and one year major acute cardiovascular events (MACE)
length of hospitalization
one year and total survival and freedom from MACE
one year target vessel failure (TVF).

CONTACTS AND LOCATIONS:
Overall Officials: Pawel E Buszman, Prof, Principal Investigator — Silesian Medical School, Poland; Stefan R Kiesz, Prof, Principal Investigator — 2San Antonio Endovascular and Heart Institute and University of Texas Health Science Center at San Antonio, Tx, USA,
Locations (5):
- United States (2):
  - Sharpe-Strumia Research Foundation of the Bryn Mawr Hospital, Bryn Mawr, PA, USA and Thomas Jefferson University, Philadelphia, Bryn Mawr, Pennsylvania
  - San Antonio Endovascular and Heart Institute and University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Poland (3):
  - Jagiellonian University, Krakow, Lesser Poland Voivodeship
  - Silesian Medical School 1-st Department of Cardiosurgery, Katowice, Silesian Voivodeship
  - Silesian Medical School 3-rd Department of Cardiology, Coronary Care Unit, Katowice, Silesian Voivodeship

REFERENCES:
- [Background] Chieffo A, Colombo A. Treatment of unprotected left main coronary artery disease with drug-eluting stents: is it time for a randomized trial? Nat Clin Pract Cardiovasc Med. 2005 Aug;2(8):396-400. doi: 10.1038/ncpcardio0272. PMID 16119701
- [Background] Chieffo A, Stankovic G, Bonizzoni E, Tsagalou E, Iakovou I, Montorfano M, Airoldi F, Michev I, Sangiorgi MG, Carlino M, Vitrella G, Colombo A. Early and mid-term results of drug-eluting stent implantation in unprotected left main. Circulation. 2005 Feb 15;111(6):791-5. doi: 10.1161/01.CIR.0000155256.88940.F8. Epub 2005 Feb 7. PMID 15699254
- [Background] Park SJ, Kim YH, Lee BK, Lee SW, Lee CW, Hong MK, Kim JJ, Mintz GS, Park SW. Sirolimus-eluting stent implantation for unprotected left main coronary artery stenosis: comparison with bare metal stent implantation. J Am Coll Cardiol. 2005 Feb 1;45(3):351-6. doi: 10.1016/j.jacc.2004.10.039. PMID 15680711
- [Background] Valgimigli M, van Mieghem CA, Ong AT, Aoki J, Granillo GA, McFadden EP, Kappetein AP, de Feyter PJ, Smits PC, Regar E, Van der Giessen WJ, Sianos G, de Jaegere P, Van Domburg RT, Serruys PW. Short- and long-term clinical outcome after drug-eluting stent implantation for the percutaneous treatment of left main coronary artery disease: insights from the Rapamycin-Eluting and Taxus Stent Evaluated At Rotterdam Cardiology Hospital registries (RESEARCH and T-SEARCH). Circulation. 2005 Mar 22;111(11):1383-9. doi: 10.1161/01.CIR.0000158486.20865.8B. PMID 15781749
- [Result] Peszek-Przybyla E, Buszman P, Bialkowska B, Zurakowski L, Banasiewicz-Szkrobka I, Debinski M, Tendera M. Stent implantation for the unprotected left main coronary artery. The long-term outcome of 62 patients. Kardiol Pol. 2006 Jan;64(1):1-6; discussion 7. PMID 16444619
- [Derived] Buszman PE, Kiesz SR, Bochenek A, Peszek-Przybyla E, Szkrobka I, Debinski M, Bialkowska B, Dudek D, Gruszka A, Zurakowski A, Milewski K, Wilczynski M, Rzeszutko L, Buszman P, Szymszal J, Martin JL, Tendera M. Acute and late outcomes of unprotected left main stenting in comparison with surgical revascularization. J Am Coll Cardiol. 2008 Feb 5;51(5):538-45. doi: 10.1016/j.jacc.2007.09.054. PMID 18237682